CLINICAL TRIAL: NCT07168096
Title: NEOPSYCO STUDY: Trajectories of Anxiety and Depression in Cancer Patients, Risk and Predictive Factors and Supportive Care; Prognostic Awareness and Shared Decision Making.
Brief Title: Trajectories of Anxiety and Depression in Cancer Patients, Risk and Predictive Factors and Supportive Care; Prognostic Awareness and Shared Decision Making.
Status: Recruiting | Type: Observational
Sponsor: Fundación Sociedad Española de Oncologia Médica (Other)
Responsible Party: Sponsor
Other Study IDs: SEOM-NEOpsico-2024-01
Record Dates: First submitted 2025-07-08; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Depression; Cancer; Anxiety
Keywords: anxiety; cancer; depression; quality of life; cognitive difficulties
MeSH Terms: conditions — Depression; Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with baseline symptoms: Patients presenting symptoms of anxiety and/or depression at the time of study inclusion. These patients will be followed to evaluate the evolution of symptoms and the impact of clinical and psychosocial variables over time
  Interventions: Other: Psychosocial and clinical assessment
- Patients without baseline symptoms: Patients without symptoms of anxiety or depression at the time of study inclusion. These participants serve as a comparison group to explore predictors of psychological distress trajectories and use of supportive care resources.
  Interventions: Other: Psychosocial and clinical assessment

INTERVENTIONS:
Other: Psychosocial and clinical assessment — Participants complete standardized self-report questionnaires and undergo medical record review at three time points (baseline, 3 months, and 6 months) to assess psychological symptoms (anxiety, depression, somatization), coping strategies, quality of life, cognitive difficulties, physical activity, nutrition, supportive care needs, and informed decision-making in the context of cancer treatment. No experimental treatment or therapy is administered.

SUMMARY:
To examine the trajectories of anxiety and depression symptoms over the course of oncological disease, and to assess potential predictors-sociodemographic (age, sex, marital status, employment status), clinical (tumor location, stage, treatment type, general health), psychological (coping strategies, quality of life, cognitive difficulties, fear of recurrence), and physical activity-and their association with support needs and utilization of psychosocial services.

DETAILED DESCRIPTION:
The study population consists of consecutive oncology patients recruited across multiple centers, with data collection occurring at baseline (diagnosis or treatment initiation) and at 3-month and 6-month follow-up time points.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of solid cancer (non-hematologic) at any stage.
* Adult age (>18 years).
* Candidate for perioperative systemic antineoplastic treatment or for advanced disease.
* Willingness to participate in the study and sign the informed consent form, as appropriate, before initiating any study-specific procedures, in accordance with good clinical practice requirements and local regulations.

Exclusion Criteria:

* Presence of a pre-existing psychiatric or neurodegenerative disorder that impairs the patient's ability to participate in the study.
* Presence of reading and writing difficulties that prevent the patient from completing the assessments.
* Receipt of oncological treatment in the past 2 years for another cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult oncology patients diagnosed with solid (non-hematologic) cancer at any stage, aged 18 years or older, who are candidates for perioperative systemic antineoplastic treatment or have advanced disease.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depression symptoms | At the time of diagnosis or treatment initiation. Follow-up at 3 months: To assess the early evolution of symptoms. Follow-up at 6 months: To analyze the medium-term evolution.
  The primary outcome of our study is psychological distress, specifically anxiety and depression symptoms, which will be measured using the Brief Symptom Inventory-18 (BSI-18).
  BSI-18 provides a single outcome measure for distress. The scoring ranges are as follows: 0-66 (low risk of depression and/or anxiety), 67-71 (intermediate risk), and >71 (clinically significant distress).

CONTACTS AND LOCATIONS:
Overall Officials: Paula Dra. Jiménez Fonseca, MD-PhD, Principal Investigator — Sociedad Española de Oncología Médica (SEOM)
Locations (18):
- Spain (18):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Ciudad Real
  - Hospital Universitario Virgen de la Luz, Cuenca, Cuenca
  - Hospital General Universitario de Elche, Alicante, Elche
  - Hospital Universitario del Sureste, Arganda, Madrid
  - Hospital Universitario La Paz, Fuencarral-El Pardo, Madrid
  - Hospital Universitario Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de La Princesa, Salamanca, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Universitario Infanta Leonor, Vallecas, Madrid
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Orense, Ourense, Orense
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz De Tenerife
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza